CLINICAL TRIAL: NCT07098975
Title: Statin Intervention for Severe Early-Onset Placental Insufficiency: A Randomized Controlled Trial Assessing Daily Administration as a Treatment Strategy (STATIN-PRE Trial)
Brief Title: Statin Intervention for Severe Early-Onset Placental Insufficiency. (STATIN-PRE Trial)
Acronym: STATIN-PRE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Universitat Autonoma de Barcelona (Other); Hospital Clinic of Barcelona (Other); Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IIBSP-PRE-2024-198
Record Dates: First submitted 2025-07-14; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Preeclampsia (PE); Intrauterine Growth Restriction (IUGR); Placental Insufficiency
Keywords: Preeclampsia; Intrauterine growth restriction; Placental Insufficiency; statins; Pravastatin
MeSH Terms: conditions — Pre-Eclampsia; Fetal Growth Retardation; Placental Insufficiency | interventions — Pravastatin

STUDY DESIGN:
Intervention Model Description: INCLUSION CRITERIA:
  * Singleton fetus.
  * Between 24+0 to 29+6 weeks of gestation at the inclusion.
  * Early-onset severe PE: women with a diagnosis of severe-preterm PE who are candidates for expectant management and have no clinical indication for immediate delivery, based on the clinical assessments of the attending doctors.
  And/or
  * IUGR: Diagnosis of early onset IUGR according to the SMFM classification with umbilical artery Doppler with absent/reversed diastolic flow; or estimated fetal weight <10th percentile plus pulsatility index (PI) of umbilical artery Doppler >95th percentil.
  * Able to give informed consent.
  EXCLUSION CRITERIA:
  * Established maternal or fetal compromise that necessitated immediate delivery
  * Abnormal karyotype, structural abnormalities, or congenital infections.
  * Treatment with pravastatin or other statins prior to inclusion
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 40mg of pravastatin (Experimental): 40 mg of pravastatin (2 pills of 20 mg at bedtime) from inclusion to delivery (estimated median of 4 weeks, maximum of 10 weeks).
  Interventions: Drug: Pravastatin 40 mg
- Placebo (Placebo Comparator): placebo of the same presentation as the active drug from inclusion to delivery (estimated median of 4 weeks, maximum of 10 weeks).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Pravastatin 40 mg — This study proposes administering a daily dose of 40 mg of pravastatin between 24 and 29.6 weeks of gestation to mothers diagnosed with preeclampsia and/or fetal growth restriction.
  Arms: 40mg of pravastatin
Other: Placebo — A visually identical but inactive pill (a placebo),
  Arms: Placebo

SUMMARY:
In pregnancies with placental insufficiency, the only available treatment is close monitoring to determine the point at which the risks of preterm birth for the baby are lower than the risks of continuing the pregnancy. Therefore, safely prolonging pregnancy is the current management goal for this condition.

Statins, such as pravastatin, are approved and marketed drugs used to prevent cardiovascular disease. Recent studies suggest that statins may help treat pregnancy complications and prolong pregnancy, thereby avoiding extreme prematurity and improving long-term health outcomes for both mother and baby.

Previous clinical trials have shown the ability of statins to stabilize angiogenic factors, thus reducing obstetric complications associated with placental insufficiency. In 2015, a study reported that pravastatin was effective in stabilizing blood pressure and reducing proteinuria associated with preeclampsia. More recently, in 2020, it was demonstrated that in pregnant women with fetal growth restriction treated with pravastatin, the sFlt-1/PlGF ratio was lower than in untreated women, indicating a slower progression of placental insufficiency.

This study proposes administering a daily dose of 40 mg of pravastatin between 24 and 29.6 weeks of gestation to mothers diagnosed with preeclampsia and/or fetal growth restriction. One group of women will receive the medication, while another group will receive a visually identical but inactive pill (a placebo), allowing us to determine whether any observed improvement in pregnancy is attributable to the medication. Assignment to the treatment or placebo group will be random, and neither the mothers nor the healthcare professionals caring for them will know which group they are in.

The investigators also aim to examine whether this intervention during pregnancy protects the cardiovascular system. For this reason, the investigators will assess both the mother and the baby six months after birth using an ultrasound of the heart and blood vessels, and the investigators will also perform a blood test on the mothers. Additionally, the investigators want to explore the needs and expectations of women who experience these complications during pregnancy and postpartum, so that their stories can guide us in finding answers and solutions that are as personalized as possible to the real needs of families. After the visit at six months postpartum, yhe investigators will follow up with annual phone calls over the next four years to check on the participants' health and their baby's. During each call, the investigators will review the participant's health status and talk about how the participant is feeling. All of this will help us ensure that the treatment does not cause any long-term issues and will improve future care for other mothers and babies.

A total of 154 pregnant women are expected to be included in order to meet the study's objectives.

DETAILED DESCRIPTION:
Preeclampsia (PE) and intrauterine growth restriction (IUGR) arise as clinical manifestations of placental insufficiency. While significant strides have been made in the prevention of PE over the past decade, resulting in a noteworthy decline in its prevalence, both PE and IUGR persist as prominent contributors to peripartum morbidity, major causes of prematurity, and sources of neonatal complications and mortality. In severe instances of PE, the potential for serious complications extends throughout pregnancy and the postpartum period, and both entities have implications on long-term maternal and children cardiovascular risks in later life.

Despite the efforts to generate successful therapeutic strategies aimed to prolong pregnancy and attenuate prematurity-related morbidity, presently, the only effective cure is timely delivery, and pharmacological therapy aims to mitigate tertiary complications such as eclampsia or severe hypertension. PE and IUGR are considered orphan diseases by the European Medicines Agency. Therefore, there is an urgent need to investigate novel drugs aimed to improve maternal and neonatal outcomes and mitigate long term sequels. Between 24 and 28 weeks of pregnancy, every day of prolongation of the pregnancy is followed by a 1-2% reduction of neonatal mortality or severe morbidity.

HMG-CoA reductase inhibitors (HMG-CoA-RI), beyond their lipid-lowering effects, have been shown to improve endothelial function, placental perfusion, have anti-inflammatory and anti-oxidant effects, and up-regulation of angiogenesis with their "pleiotropic effects". These HMG-CoA-RI related beneficial properties suggest their potential protective potential during the acute phase of placental insufficiency and subsequent protection on cardiovascular maternal and fetal programming.

It is our WORKING HYPOTHESIS that 40 mgr of oral administration of pravastatin daily will prolong duration of pregnancy and will provide cardioprotection and additional benefits to both mother and neonates to that afforded by conventional management of PE and IUGR.

FIRST AIM: To assess that daily 40 mgr of oral administration of pravastatin in pregnant individuals with PE and/or IUGR between 24.0 and 29.6 weeks of gestation will prolong duration of pregnancy compared to conventional management.

SECOND AIM: Determine whether pravastatin improve cardiac function, placental perfusion, angiogenesis, total antioxidant status (TAS) and lipid profile during pregnancy and after pregnancy in both mothers and neonates in the intervention group compared to controls.

THIRD AIM: To evaluate changes in genetic expression profile in human tissues after treatment with novel statins' therapy.

FOURTH AIM: To include women's needs and expectations about PE, IUGR and preterm birth and future heath in order to improve the success of the translation into real changes in women and infant health.

ELIGIBILITY:
Inclusion Criteria:

* Singleton fetus.
* Between 24+0 to 29+6 weeks of gestation at the inclusion.
* Early-onset severe PE: women with a diagnosis of severe-preterm PE who are candidates for expectant management and have no clinical indication for immediate delivery, based on the clinical assessments of the attending doctors.

And/or

* IUGR: Diagnosis of early onset IUGR according to the SMFM classification with umbilical artery Doppler with absent/reversed diastolic flow; or estimated fetal weight <10th percentile plus pulsatility index (PI) of umbilical artery Doppler >95th percentil.
* Able to give informed consent.

Exclusion Criteria:

* Established maternal or fetal compromise that necessitated immediate delivery
* Abnormal karyotype, structural abnormalities, or congenital infections.
* Treatment with pravastatin or other statins prior to inclusion.
* Lactose intolerance

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Days of prolongation of pregnancy between inclusion and delivery. | From date of randomization until the date of delivery, assesed up to 10 weeks

SECONDARY OUTCOMES:
Maternal pregnancy-related morbidity composite score | At delivery
  Including any of the following:
  (i) HELLP syndrome .(ii)Central nervous system dysfunction (iii)Hepatic dysfunction (iv) renal dysfunction . (v)Respiratory dysfunction. (vi)Cardiovascular dysfunction. (vii) Placental abruption. (viii) a requirement for transfusion of blood products red cells, platelets, fresh frozen plasma and cryoprecipitate. Minimum score of 0, maximum score of 8. Higher scores mean worse outcome.
Preterm birth before 34 weeks of gestation | At delivery
Birth weight | At delivery
Neonatal acidosis | At delivery
  arterial pH <7.10+ base excess >12 mEq/L
Perinatal mortality | from 22 weeks of gestation to 28 days post-partum
Days in the neonatal intensive care | From date of delivery until the date of discharge of the neonatal intensive care or date of death from any cause, whichever came first, assessed up to 3 months
Neonatal morbidity | At delivery
Maternal/ fetal cardiac function | at inclusion, at delivery and at 6 months after delivery
  In the echocardiographic ultrasound assessment at inclusion, at delivery and at 6 months after delivery
Biomarkers in maternal blood | at the time of diagnosis and delivery
  soluble fms-like tyrosine kinase 1 (sFlt1) and placental growth factor (PlGF); NTProBNP, continuous (pg/mL)
Biomarkers in umbilical cord blood | At delivery
  sFlt1, PlGF and NTProBNP
Concentrations in plasma/serum | Since inlcusion until 6 months after delivery
  of dense low density lipoprotein (dense LDL), apolipoprotein CIII (apoCIII), and TAS
Increased cardiovascular risk by blood preassure measurement, echocardiographic assessment, global longitudinal strain, carotid-ntima-media thickness, Ophtalmic artery Doppler evaluation, IBERLIFERISK score. | 6 months after delivery
  Defined by any of the following (binary(yes/no): (1)Presence of hypertension, defined as stage 1 hypertension (SBP of 130-139 or DBP of 80-89 mmHg) and/or (2)Proteinuria>300 mg/24 hours or renal insufficiency and/or (3)High-risk CVD according to IBERLIFERISK score (score >50%) and/or (4) IMT >p90 according to the Spanish population (5) Abnormal cardiac function in the echocardiographic ultrasound assessment. Abnormal values of the different parameters will be considered according to reference limits in pregnancy and post-partum published in 2023 by the British Society of Echocardiography and/or (6) Abnormal biochemical cardiac markers (NTproBNP, high-sensitivity troponin) and/or (7) Cardiovascular major events (ictus, coronary artery disease, cardiac insufficiency or myocardiopathy).
Cardiovascular algorithms and cloud-based analysis and decision support system | Through study completion, an avarage of 4 years
  Initially, we will aggregate patient data from diverse sources like electronic health records, medical imaging, biochemical and lipid results forming a comprehensive patient profile. This data undergoes feature extraction and preprocessing to identify relevant parameters and ensure consistency.
  We will develop an algorithm, incorporating machine learning techniques. This algorithm will be of use to predict cardiovascular risks in women after a placental complication. The computational demands are met through the utilization of cloud infrastructure, providing secure storage and real-time processing capabilities. The results generated by this algorithm will be integrated into user-friendly interfaces, forming a decision support system for healthcare professionals. This assists them in making well-informed decisions regarding patient care, treatment plans, and interventions.
mRNAs in trophoblast | At delivery
  Gene expression of: IL-6, IFN-γ, TNF-α, VEGFA, VEGFB, FGF2, and RQVEGF Receptor1

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital de la Santa Creu i de Sant Pau, Barcelona, barcelona
  - Hospital Clínic de Barcelona, Barcelona, Barcelona

IPD SHARING:
Plan to Share IPD: Yes
Aligned with open science principles and Horizon Europe guidelines, our project prioritizes transparency and reproducibility. Data will be openly shared on the Open Science Framework (OSF), guided by FAIT principles for accessibility and reusability. Biobanked samples will be accessible to other researchers, fostering collaboration and further exploration.